CLINICAL TRIAL: NCT03492216
Title: Drinkers' Intervention to Prevent Tuberculosis (DIPT Study)
Acronym: DIPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Infectious Diseases Research Collaboration, Uganda (Other); Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 17-22727
Record Dates: First submitted 2018-02-20; First posted 2018-04-10 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: HIV/AIDS; Tuberculosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): All participants will receive brief alcohol and adherence counseling according to Uganda Ministry of Health guidelines.
- Escalating incentives (EtG tests) (Experimental): Escalating incentives for EtG negative urine test (Intervention: Incentives for negative EtG test).
  Interventions: Behavioral: Incentives for negative EtG test
- Escalating incentives (IsoScreen tests) (Experimental): Escalating incentives for IsoScreen positive urine tests (Intervention: Incentives for positive IsoScreen test).
  Interventions: Behavioral: Incentives for positive IsoScreen test
- Escalating incentives (EtG + IsoScreen) (Experimental): Escalating incentives for EtG negative tests and for IsoScreen positive urine tests with the incentives rewarded separately (Interventions: Incentives for negative EtG test and Incentives for positive IsoScreen test).
  Interventions: Behavioral: Incentives for negative EtG test; Behavioral: Incentives for positive IsoScreen test

INTERVENTIONS:
Behavioral: Incentives for negative EtG test — Economic incentives are given to the study participant contingent on point-of-care (POC) urine ethyl glucuronide (EtG) <300 ng/mL with the amount of the incentive escalating with each subsequent negative EtG test.
  Arms: Escalating incentives (EtG + IsoScreen); Escalating incentives (EtG tests)
Behavioral: Incentives for positive IsoScreen test — Economic incentives contingent on POC (IsoScreen) INH urine positive tests with the amount of the incentive escalating with each subsequent positive IsoScreen test.
  Arms: Escalating incentives (EtG + IsoScreen); Escalating incentives (IsoScreen tests)

SUMMARY:
There is an urgent global need to decrease the high mortality of tuberculosis (TB) in persons with HIV as TB is the leading cause of death among persons with HIV worldwide. The DIPT (Drinkers' Intervention to Prevent TB) study is a randomized, 2x2 factorial trial among HIV/TB co-infected adults in Uganda with heavy alcohol use (n=680 persons, 340 each U01). The goal of the study is to determine whether economic incentive interventions can promote both reduced alcohol use and isoniazid (INH) pill taking among HIV/TB co-infected adult heavy drinkers, during isoniazid preventive therapy (IPT: a six-month course of INH) at HIV clinics in southwestern Uganda. Participants will be randomized to one of four arms: Arm 1: no incentives (control); Arm 2: economic incentives for decreasing alcohol use only; Arm 3: economic incentives for IPT adherence only; Arm 4: economic incentives for decreasing alcohol use and for IPT adherence (rewarded independently).

DETAILED DESCRIPTION:
TB is the leading cause of death among persons with HIV worldwide, and HIV-infected drinkers are at very high risk for TB disease and mortality. Globally, an estimated 25% of persons with HIV are heavy drinkers, and the risk of TB disease is 3-fold higher among heavy drinkers compared to non-drinkers. Six months of isoniazid (INH) preventive therapy (IPT) reduces TB morbidity and mortality by 30-50% above the benefit of antiretroviral therapy (ART). However, INH can be toxic to the liver, and as a result in many high TB/HIV prevalence settings, such as east Africa, heavy drinkers are not offered IPT. Thus interventions to reduce alcohol use are needed to decrease INH toxicity during IPT among HIV/TB infected drinkers. It is also well established that heavy drinkers have poorer ART adherence, and there is growing evidence of reduced IPT adherence in drinkers. However, interventions to reduce drinking have had limited impact on ART adherence, and further interventions to increase IPT adherence among HIV/TB infected drinkers are likely needed.

The use of incentives to promote healthy behavior is a highly effective approach for reducing substance use and for improving adherence to HIV and TB regimens in resource-rich settings. Economic incentives to reduce alcohol use may create a window for safe and effective IPT use over six months by decreasing hepatotoxicity. Decreases in alcohol use may also improve IPT adherence, or additional incentives for IPT adherence may be needed. Such strategies to reduce alcohol use have not been studied in low-income countries and the effectiveness of incentives to optimize IPT in HIV/TB co-infected drinkers is unknown.

OBJECTIVES

Aim 1: Alcohol Reduction Intervention: Determine the effectiveness of economic incentives contingent on point-of-care (POC) urine ethyl glucuronide (EtG) <300 ng/mL (Arms 2 & 4) versus no alcohol incentives (Arms 1 & 3) to reduce heavy drinking over 6 months, among HIV/TB co-infected adult drinkers receiving IPT. The investigators will randomize participants to low-cost escalating prize incentives for EtG negative urine tests at IPT refill visits (Arms 2+4), versus no incentives (Arms 1+3).

Aim 2: INH Adherence Intervention: Determine the effectiveness of economic incentives contingent on POC (IsoScreen) INH urine positive tests (Arms 3 & 4) versus no INH incentives (Arms 1 & 2) on INH adherence among HIV/TB co-infected adult drinkers. The investigators will randomize participants to low-cost escalating prize incentives for INH positive urine tests at IPT refill visits (Arms 3+4), versus no incentives (Arms 1+2).

Aim 3: Impact Assessment of Intervention: Assess the impact of economic incentives on HIV virologic suppression and explore their mechanisms of action, six months after trial completion. The investigators will follow all study participants for six months after trial completion.

1. Assess the impact of the 3 separate incentive interventions (Arms 2, 3, 4) vs. no incentives (Arm 1) on HIV virologic suppression.
2. Explore the mechanisms that may drive the economic incentives to increase virologic suppression. Potential mediators will be reductions in alcohol use and level of IPT adherence.

This study will leverage new low-cost POC tests for alcohol use and INH pill-taking for the first study of incentive-based alcohol and adherence interventions in low-resource settings; these interventions may improve the safety and effectiveness of life-saving medications for heavy alcohol users in many settings.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected adult (≥18 years) prescribed antiretroviral therapy (ART) for at least 6 months;
* Current heavy alcohol use (AUDIT-C positive for prior 3 month drinking and positive EtG urine test);
* Positive tuberculin skin test (TST) (≥5 mm induration);
* AST and ALT <2x the upper limit of normal (ULN);
* Fluent in Runyankole or English;
* No history of active TB, TB treatment, or TB preventive therapy;
* Lives within 2-hour travel time or 60 km of the study site.

Exclusion Criteria:

* Prescribed nevirapine (NVP, an ART drug that is declining in usage due to high risk for hepatotoxicity);
* Plans to move out of the catchment area within 6 months;
* Prescribed anti-convulsion medications or history of recurring seizures;
* ALT or AST elevations (>2X ULN);
* Suspected or confirmed active TB as determined by symptom screening and followed by chest X-ray and sputum testing;
* History of prior active TB treatment or prior IPT.
* Pregnant at time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Hahn, PhD, Principal Investigator — University of California, San Francisco; Gabriel Chamie, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- Uganda (2):
  - Infectious Disease Research Collaboration (IDRC), Mbarara
  - Mbarara Regional Referral Hospital (MRRH): Immune Suppression Syndrome HIV, Mbarara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muyindike WR, Fatch R, Lodi S, Emenyonu NI, Kekibiina A, Adong J, Beesiga B, Marson K, Thirumurthy H, McDonell MG, Kamya MR, Chamie G, Hahn JA. Alcohol use and HIV suppression after completion of financial incentives for alcohol abstinence and isoniazid adherence: a randomized controlled trial. EClinicalMedicine. 2025 Jan 8;80:103045. doi: 10.1016/j.eclinm.2024.103045. eCollection 2025 Feb. PMID 39867970
- [Derived] Chamie G, Hahn JA, Kekibiina A, Emenyonu NI, Beesiga B, Marson K, Fatch R, Lodi S, Adong J, Thirumurthy H, McDonell MG, Gandhi M, Bryant K, Havlir DV, Kamya MR, Muyindike WR. Financial incentives for reduced alcohol use and increased isoniazid adherence during tuberculosis preventive therapy among people with HIV in Uganda: an open-label, factorial randomised controlled trial. Lancet Glob Health. 2023 Dec;11(12):e1899-e1910. doi: 10.1016/S2214-109X(23)00436-9. PMID 37973340
- [Derived] Lodi S, Emenyonu NI, Marson K, Kwarisiima D, Fatch R, McDonell MG, Cheng DM, Thirumurthy H, Gandhi M, Camlin CS, Muyindike WR, Hahn JA, Chamie G. The Drinkers' Intervention to Prevent Tuberculosis (DIPT) trial among heavy drinkers living with HIV in Uganda: study protocol of a 2x2 factorial trial. Trials. 2021 May 20;22(1):355. doi: 10.1186/s13063-021-05304-7. PMID 34016158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment occurred from April 2018 through July 2021. 5,508 persons were screened and 680 persons were enrolled and randomized.
Groups:
- Escalating Incentives (Ethyl Glucuronide [EtG] Tests): Escalating incentives for ethyl glucuronide (EtG) negative urine test (Intervention: Incentives for negative EtG test).
  Incentives for negative EtG test: Economic incentives are given to the study participant contingent on point-of-care (POC) urine EtG <300 ng/mL with the amount of the incentive escalating with each subsequent negative EtG test.
- Escalating Incentives (IsoScreen Tests): Escalating incentives for IsoScreen positive urine tests (Intervention: Incentives for positive IsoScreen test).
  Incentives for positive IsoScreen test: Economic incentives contingent on point-of-care IsoScreen (Isoniazid, INH) urine positive tests with the amount of the incentive escalating with each subsequent positive IsoScreen test.
- Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen): Escalating incentives for ethyl glucuronide (EtG) negative tests and for IsoScreen positive urine tests, with the incentives rewarded separately (Interventions: Incentives for negative EtG test and Incentives for positive IsoScreen test).
  Incentives for negative EtG test: Economic incentives are given to the study participant contingent on point-of-care (POC) urine ethyl glucuronide (EtG) <300 ng/mL with the amount of the incentive escalating with each subsequent negative EtG test.
  Incentives for positive IsoScreen test: Economic incentives contingent on POC (IsoScreen) INH urine positive tests with the amount of the incentive escalating with each subsequent positive IsoScreen test.
Period: Overall Study
Arm/Group | Control | Escalating Incentives (Ethyl Glucuronide [EtG] Tests) | Escalating Incentives (IsoScreen Tests) | Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen)
Started | 169 | 169 | 170 | 172
3 Month Visit | 158 | 162 | 166 | 168
6 Month Visit | 154 | 164 | 162 | 165
Completed (Completed 12-month follow-up visit) | 149 | 160 | 153 | 158
Not Completed | 20 | 9 | 17 | 14
Not completed — Death | 1 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 5 | 3 | 1 | 1
Not completed — Lost to Follow-up | 9 | 2 | 7 | 8
Not completed — Moved | 5 | 3 | 3 | 5
Not completed — Too ill | 0 | 1 | 0 | 0
Not completed — Incarcerated | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Escalating Incentives (Ethyl Glucuronide [EtG] Tests): Escalating incentives for ethyl glucuronide (EtG) negative urine test (Intervention: Incentives for negative EtG test).
  Incentives for negative EtG test: Economic incentives are given to the study participant contingent on point-of-care urine EtG <300 ng/mL with the amount of the incentive escalating with each subsequent negative EtG test.
- Escalating Incentives (IsoScreen Tests): Escalating incentives for IsoScreen positive urine tests (Intervention: Incentives for positive IsoScreen test).
  Incentives for positive IsoScreen test: Economic incentives contingent on point-of-care IsoScreen (Isnoiazid, INH) urine positive tests with the amount of the incentive escalating with each subsequent positive IsoScreen test.
- Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen): Escalating incentives for ethyl glucuronide (EtG) negative tests and for IsoScreen positive urine tests with the incentives rewarded separately (Interventions: Incentives for negative EtG test and Incentives for positive IsoScreen test).
  Incentives for negative EtG test: Economic incentives are given to the study participant contingent on point-of-care (POC) urine EtG <300 ng/mL with the amount of the incentive escalating with each subsequent negative EtG test.
  Incentives for positive IsoScreen test: Economic incentives contingent on POC (IsoScreen) INH urine positive tests with the amount of the incentive escalating with each subsequent positive IsoScreen test.
- Total: Total of all reporting groups
Arm/Group | Control | Escalating Incentives (Ethyl Glucuronide [EtG] Tests) | Escalating Incentives (IsoScreen Tests) | Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen) | Total
Number analyzed (Participants) | 169 | 169 | 170 | 172 | 680
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 167 | 164 | 167 | 169 | 667
  >=65 years | 2 | 5 | 3 | 3 | 13
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [33 to 46] | 38 [32 to 46] | 40 [32 to 48] | 39 [31 to 46] | 39 [32 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 53 | 53 | 53 | 210
  Male | 118 | 116 | 117 | 119 | 470
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Uganda | 169 | 169 | 170 | 172 | 680

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With and Without Non-hazardous Drinking, as Determined by Self-report and the Biomarker Phosphatidylethanol, at 3- and 6-months.
Description: Non-hazardous drinking is a composite outcome, measured at both 3 and 6 months. An individual must meet criteria for non-hazardous drinking (Alcohol Use Disorders Identification Test - Consumption [AUDIT-C], prior 3 months, negative) and phosphatidylethanol (PEth) <35 ng/mL) at both time-points (3- and 6-months) in order to achieve the outcome.
Time Frame: Both 3 months and 6 months (composite measure)
Population: As pre-specified in the Study Protocol, participants in the EtG incentive arms (2 + 4) were compared to those in the no EtG incentive arms (1 + 3).
  EtG incentives (arms 2 + 4): 323/341 participants included; 18/341 participants excluded.
  No EtG incentives (arms 1 + 3): 313/339 participants included; 26/339 participants excluded.
Measure: Count of Participants; unit: Participants
Groups:
- Alcohol Incentives: Escalating incentives for ethyl glucuronide (EtG) negative urine test (Intervention: Incentives for negative EtG test). (Arms 2 + 4)
- No Alcohol Incentives: No ethylglucuronide (EtG) testing; no incentives for EtG negative urine test. (Arms 1 + 3)
Arm/Group | Alcohol Incentives | No Alcohol Incentives
Number analyzed (Participants) | 323 | 313
Participants
  Non-hazardous alcohol use at 3 and 6 months = yes | 57 | 31
  Non-hazardous alcohol use at 3 and 6 months = no | 266 | 282
Statistical Analysis 1: Comparison: Alcohol Incentives vs No Alcohol Incentives; Test type: Superiority; p = 0.0025, Regression, Logistic; Risk Difference (RD) = 7.6, 95% CI 2-sided [2.7 to 12.5] — adjusted risk difference for non-hazardous alcohol use, alcohol incentive groups compared to no alcohol incentive groups. logistic regression model adjusted for INH incentive arm, participant sex, and study site

2. Primary Outcome: Number of Participants With >90% Isoniazid (INH) Adherence During Prescribed Course of INH
Description: Isoniazid (INH) adherence percentage is defined as the number of days with >0 pill bottle openings divided by the number of prescribed doses, times 100. Pill bottle openings are captured by the Medication Event Monitoring System (MEMS) pill cap, with no more than 1 opening per day counted. The INH adherence outcome is INH adherence percentage, dichotomized as >90% versus <= 90%.
Time Frame: 6 months
Population: As pre-specified in the Study Protocol, participants in the INH incentive arms (3 + 4) were compared to those in the no INH incentive arms (1 + 2).
  INH incentive group (arms 3 + 4): 335/342 participants are included; 7 are excluded.
  No INH incentive group (arms 1 + 2): 321/338 participants are included; 17 are excluded.
Measure: Count of Participants; unit: Participants
Groups:
- Isoniazid (INH) Adherence Incentives: Escalating incentives for IsoScreen positive INH urine tests (Intervention: Incentives for positive IsoScreen test).
- No Incentives for Isoniazid (INH) Adherence: No IsoScreen INH urine tests (no incentives for INH adherence).
Arm/Group | Isoniazid (INH) Adherence Incentives | No Incentives for Isoniazid (INH) Adherence
Number analyzed (Participants) | 335 | 321
Participants
  >90% INH adherence | 244 | 234
  <=90% INH adherence | 91 | 87
Statistical Analysis 1: Comparison: Isoniazid (INH) Adherence Incentives vs No Incentives for Isoniazid (INH) Adherence; Test type: Superiority; p = 0.9435, Regression, Logistic; Risk Difference (RD) = -0.2, 95% CI 2-sided [-7.0 to 6.5] — adjusted risk difference for >90% INH adherence, INH incentive group compared to no INH incentives. logistic regression model adjusted for alcohol incentive arm, participant sex and study site

3. Secondary Outcome: Number of Participants With Hepatotoxicity Resulting in Isoniazid (INH) Discontinuation.
Description: Isoniazid (INH) treatment discontinuation due to a Grade 3+ hepatotoxicity at any time during the treatment period. Grade 3 hepatoxicity is defined by lab and/or clinical criteria as alanine transaminase (ALT) or aspartate transaminase (AST) elevation ≥5 (but <10) times the upper limit of normal and/or symptoms consistent with hepatotoxicity; and Grade 4 as ALT or AST elevation ≥10 times the upper limit of normal or potentially life-threatening symptoms.
Time Frame: up to 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Escalating Incentives (Ethyl Glucuronide [EtG] Tests): Escalating incentives for ethyl glucuronide (EtG) negative urine test (Intervention: Incentives for negative EtG test).
  Incentives for negative EtG test: Economic incentives are given to the study participant contingent on point-of-care urine EtG) <300 ng/mL with the amount of the incentive escalating with each subsequent negative EtG test.
- Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen): Escalating incentives for ethyl glucuronide (EtG) negative tests and for IsoScreen positive urine tests with the incentives rewarded separately (Interventions: Incentives for negative EtG test and Incentives for positive IsoScreen test).
  Incentives for negative EtG test: Economic incentives are given to the study participant contingent on point-of-care (POC) urine EtG <300 ng/mL with the amount of the incentive escalating with each subsequent negative EtG test.
  Incentives for positive IsoScreen test: Economic incentives contingent on POC IsoScreen (Inosiazid, INH) urine positive tests with the amount of the incentive escalating with each subsequent positive IsoScreen test.
Arm/Group | Control | Escalating Incentives (Ethyl Glucuronide [EtG] Tests) | Escalating Incentives (IsoScreen Tests) | Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen)
Number analyzed (Participants) | 169 | 169 | 170 | 172
Participants | 13 | 10 | 15 | 9

4. Secondary Outcome: INH Concentration in Hair
Description: Secondary Outcome. INH concentration in hair captures INH adherence over a period of weeks to months. Hair samples collected at the 3- and 6-month study visits will be analyzed for INH concentration.
Time Frame: 3 and 6 months
Population: Only participants in the INH adherence incentive arms had INH concentration in hair analyzed.
Measure: Median (Inter-Quartile Range); unit: pmol INH + AcINH / mg hair
Arm/Group | Control | Escalating Incentives (Ethyl Glucuronide [EtG] Tests) | Escalating Incentives (IsoScreen Tests) | Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen)
Number analyzed (Participants) | 0 | 0 | 150 | 153
pmol INH + AcINH / mg hair
  at 3 months: number analyzed (Participants) | 0 | 0 | 141 | 146
  at 3 months |  |  | 49.4 [26.8 to 81.3] | 49.1 [28.0 to 81.1]
  at 6 months: number analyzed (Participants) | 0 | 0 | 124 | 130
  at 6 months |  |  | 49.3 [27.4 to 78.8] | 57.1 [31.9 to 84.0]

5. Secondary Outcome: Number of Participants With and Without HIV Viral Suppression at 12 Months
Description: The percentage of study participants with HIV viral load suppression (defined as <200 copies/ml) at 12 months post-enrollment.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Escalating Incentives (Ethyl Glucuronide [EtG] Tests) | Escalating Incentives (IsoScreen Tests) | Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen)
Number analyzed (Participants) | 148 | 155 | 149 | 148
Participants
  HIV viral suppression = yes | 144 | 147 | 146 | 146
  HIV viral suppression = no | 4 | 8 | 3 | 2
Statistical Analysis 1: Comparison: Control vs Escalating Incentives (Ethyl Glucuronide [EtG] Tests); Test type: Superiority; p = 0.26, Regression, Logistic; Risk Difference (RD) = -2.5, 95% CI 2-sided [-6.8 to 1.9] — adjusted risk different for HIV viral suppression at 12 months, Arm 2 (escalating incentives; EtG tests) compared to Arm 1 (control); logistic regression model adjusted for randomization arm, participant sex, and study site
Statistical Analysis 2: Comparison: Control vs Escalating Incentives (IsoScreen Tests); Test type: Superiority; p = 0.70, Regression, Logistic; Risk Difference (RD) = 0.7, 95% CI 2-sided [-2.8 to 4.1] — adjusted risk different for HIV viral suppression at 12 months, Arm 3 (escalating incentives; IsoScreen tests) compared to Arm 1 (control); logistic regression model adjusted for randomization arm, participant sex, and study site
Statistical Analysis 3: Comparison: Control vs Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen); Test type: Superiority; p = 0.42, Regression, Logistic; Risk Difference (RD) = 1.3, 95% CI 2-sided [-1.9 to 4.5] — adjusted risk different for HIV viral suppression at 12 months, Arm 4 (escalating incentives; EtG and IsoScreen tests) compared to Arm 1 (control); logistic regression model adjusted for randomization arm, participant sex, and study site

6. Secondary Outcome: Number of Participants With Active Tuberculosis (TB).
Description: Secondary Outcome. Number of participants diagnosed with active TB, within the 12 months of study follow-up.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Escalating Incentives (Ethyl Glucuronide [EtG] Tests) | Escalating Incentives (IsoScreen Tests) | Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen)
Number analyzed (Participants) | 169 | 169 | 170 | 172
Participants | 0 | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the course of the study follow-up (1 year).
Arm/Group | Control | Escalating Incentives (Ethyl Glucuronide [EtG] Tests) | Escalating Incentives (IsoScreen Tests) | Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen)
All-Cause Mortality (participants affected / at risk) | 1/169 | 0/169 | 4/170 | 0/172
Serious Adverse Events (participants affected / at risk) | 5/169 | 5/169 | 8/170 | 4/172
Other Adverse Events (participants affected / at risk) | 64/169 | 50/169 | 55/170 | 39/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=169) | Escalating Incentives (Ethyl Glucuronide [EtG] Tests) (N=169) | Escalating Incentives (IsoScreen Tests) (N=170) | Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen) (N=172)
Physical assault; hospitalization (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Elevated ALT or AST (Hepatobiliary disorders) | 3 (3) | 2 (2) | 3 (3) | 3 (3) — Grade 4 aspartate transaminase (AST) or alanine transaminase (ALT) elevation defined as AST or ALT >=10 times the upper limit of normal (ULN).
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization; surgery for intestinal obstruction
Alcohol withdrawal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Alcohol withdrawal delirium and alcohol induced psychosis
Road traffic accident; hospitalization (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Bronchopneumonia resulting in hospitalization
Hospitalization (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hospitalization secondary to prior spontaneous abortion
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — cause unknown
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — esophageal tumor/regurgitation of food
Death (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — developed active tuberculosis
Death (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — sepsis
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Per post-mortem report, had bronchopneumonia and haemorrhagic pancreatitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=169) | Escalating Incentives (Ethyl Glucuronide [EtG] Tests) (N=169) | Escalating Incentives (IsoScreen Tests) (N=170) | Escalating Incentives (Ethyl Glucuronide [EtG] + IsoScreen) (N=172)
Grade 3: elevated AST or ALT (Hepatobiliary disorders) | 12 (12) | 7 (8) | 14 (14) | 9 (9) — Grade 3 aspartate transaminase (AST) or alanine transaminase (ALT) elevation defined as AST or ALT >=5 to < 10 times the upper limit of normal (ULN).
Grade 2: elevated AST or ALT (Hepatobiliary disorders) | 52 (66) | 42 (66) | 40 (51) | 31 (43) — Grade 2 aspartate transaminase (AST) or alanine transaminase (ALT) elevation defined as AST or ALT >2 to < 5 times the upper limit of normal (ULN).
Myalgia of thighs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia of knees (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced lupus (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Active TB (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Blurry vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Elevated creatinine (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Low platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT03492216/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT03492216/SAP_001.pdf